CLINICAL TRIAL: NCT07196696
Title: An in Vivo CT Imaging Study After Insertion of the LMA Supreme, I-gel, and GMA-Tulip Airway Devices Under General Anesthesia (GLAM-II)
Brief Title: An in Vivo CT Imaging Study of GMA-Tulip, I-gel, and LMA Supreme (GLAM-II)
Acronym: GLAM-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wang Jiangling, Principal Investigator, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: IRB-2025-1160（IIT）
Record Dates: First submitted 2025-09-21; First posted 2025-09-29 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Supraglottic Airway Device
Keywords: GMA-Tulip; I-gel; LMA-Supreme; Supraglottic airway device

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GMA-Tulip (Experimental): Insert GMA-Tulip in this group and observe the outcomes
  Interventions: Device: GMA-Tulip
- I-gel (Active Comparator): Insert I-gel in this group and observe the outcomes
  Interventions: Device: I-gel
- LMA-Supreme (Sham Comparator): Insert LMA-Supreme in this group and observe the outcomes
  Interventions: Device: LMA-Supreme insertion

INTERVENTIONS:
Device: GMA-Tulip — Under general anesthesia, GMA-Tulip laryngeal mask is inserted following standardized protocols. CT scanning and fiberoptic laryngoscopy are performed to assess insertion depth, anatomical alignment, and tissue compression.
  Other Names: GMA-Tulip insertion
  Arms: GMA-Tulip
Device: I-gel — Under general anesthesia, I-gel laryngeal mask is inserted following standardized protocols. CT scanning and fiberoptic laryngoscopy are performed to assess insertion depth, anatomical alignment, and tissue compression.
  Other Names: I-gel insertion
  Arms: I-gel
Device: LMA-Supreme insertion — Under general anesthesia, LMA Supreme laryngeal mask is inserted following standardized protocols. CT scanning and fiberoptic laryngoscopy are performed to assess insertion depth, anatomical alignment, and tissue compression.
  Other Names: LMA-Supreme
  Arms: LMA-Supreme

SUMMARY:
Laryngeal masks are core devices for supraglottic airway management, and the accuracy of their anatomical position directly impacts ventilation safety and the incidence of complications. Despite their wide clinical application, gaps remain in understanding their in vivo anatomical characteristics. This study aims to evaluate the in vivo anatomical features (e.g., insertion depth, anatomical alignment, tissue compression) of three laryngeal masks (LMA Supreme, I-gel, GMA-Tulip) using CT scanning in anesthetized patients undergoing CT interventional therapy, providing anatomical evidence for optimized laryngeal mask selection and complication prevention.

DETAILED DESCRIPTION:
After approval by the Ethics Committee of Zhejiang Cancer Hospital (Approval Number: IRB-2025-001 (IIT)), this study will be registered on ClinicalTrials.gov prior to participant enrollment. Written informed consent will be obtained from all participants. The study is planned to be conducted from September 2025 to December 2025.

Eligible participants are 18-75 years old, ASA physical status I-II, BMI <30 kg/m², scheduled for CT interventional therapy, and without contraindications (e.g., head/neck airway anomalies, participation in other clinical studies).

Pre-procedure Preparation: Patients fast and abstain from fluids as per standard protocols, with no premedication. Upon admission to the operating room, standard monitoring (ECG, HR, BP, SpO₂) is initiated, and an intravenous access is established. Pre-anesthesia baseline HR and BP are recorded.

Anesthesia Induction: Pre-oxygenation with 8 L/min oxygen via face mask for 3 minutes. Anesthesia is induced with propofol (3.5 μg/ml) and remifentanil (4 ng/ml). After loss of eyelash reflex, rocuronium (0.9 mg/kg) is administered, and laryngeal mask insertion is performed 2 minutes post-rocuronium injection.

Laryngeal Mask Insertion: Participants are randomly assigned (via computer-generated sequence) to one of three groups: LMA Supreme Group (L Group), I-gel Group (I Group), or GMA-Tulip Group (G Group). Each patient receives one laryngeal mask insertion by an anesthesiologist with ≥5 years of experience, following standardized insertion protocols for each device:

LMA Supreme: Lubricate the posterior surface; place the head in neutral or sniffing position; advance the mask along the midline of the oral cavity until resistance is felt.

I-gel: Lubricate the posterior surface; advance along the hard palate until definite resistance is felt.

GMA-Tulip: Lubricate the posterior surface; place the head in sniffing position; avoid tongue entrapment; advance until passing the base of the tongue (no need to seek strong resistance); gently shake to ensure tight fit.

Laryngeal mask size is selected based on body weight:

L Group: 3# (30-50 kg), 4# (50-70 kg), 5# (70-100 kg); I Group: 3# (30-60 kg), 4# (50-90 kg), 5# (>90 kg); G Group: 2.5# (<60 kg), 3# (60-85 kg), 4# (>80 kg);

Anesthesia Maintenance: Propofol (3.5 μg/ml) and remifentanil (2 ng/ml) are infused to maintain BIS 40-60. Additional rocuronium (0.15 mg/kg) or sufentanil (5 μg) is administered as needed. Hemodynamics are maintained within ±20% of baseline using medications (atropine, ephedrine, esmolol, dopamine, norepinephrine, nitroglycerin) if required. At the end of the procedure, propofol and remifentanil are discontinued, and rocuronium is antagonized with sugammadex sodium (200 mg). The laryngeal mask is removed when the patient regains consciousness and can follow commands. Participants recover in the Post-Anesthesia Care Unit (PACU) for ≥1 hour before discharge.

Alignment Verification: Mechanical ventilation is initiated with parameters: VT 6-8 ml/kg, I:E 1:2, RR 12-14 breaths/min, maintaining PETCO₂ 35-45 mmHg. Air tightness is confirmed via leak test (25 cmH₂O pressure) and auscultation. Fiberoptic laryngoscopy is used to grade anatomical alignment (Grade I: Only one aryepiglottic fold and partial laryngeal inlet visible, SpO₂ >98%; Grade II: Bilateral aryepiglottic folds and partial laryngeal inlet visible, SpO₂ >98%; Grade III: Bilateral aryepiglottic folds, laryngeal inlet, and partial glottis visible; Grade IV: Entire glottis visible).

Outcome Assessment: CT scanning is performed to measure insertion depth, anatomical alignment, and tissue compression. Post-procedure follow-up is conducted at 24 hours to assess complications (mucosal injury, hoarseness, sore throat via VAS 0-10, regurgitation).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years, scheduled for CT interventional therapy;
* Aged 18-75 years, scheduled for CT interventional therapy;
* Body Mass Index (BMI) <30 kg/m²;
* Good communication and cooperation, with voluntary signing of the informed consent form.

Exclusion Criteria:

* Presence of head/neck or airway anatomical abnormalities (e.g., laryngeal cartilage malformation, Grade III tonsillar hypertrophy, tongue hypertrophy, cervical spine malformation) that may affect laryngeal mask insertion or CT imaging evaluation;
* Current participation in other clinical studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-10-12 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Insertion depth of the three laryngeal masks | During CT scanning immediately after laryngeal mask insertion (within 30 minutes of insertion)
  Measurement of the distance from the laryngeal mask tip to the glottis and the upper edge of the 5th cervical vertebra (C5), and the relationship between the mask tip and the cricoid cartilage plate (via CT imaging)

SECONDARY OUTCOMES:
Anatomical alignment of the three laryngeal masks | During fiberoptic examination and CT scanning immediately after laryngeal mask insertion
  Assessment of laryngeal inlet coverage (glottis, epiglottis, aryepiglottic folds, arytenoid cartilage, interarytenoid notch) via fiberoptic laryngoscopy (graded as Grade I-IV) and CT imaging.
Degree of local tissue compression | During CT scanning immediately after laryngeal mask insertion.
  Quantification of epiglottis/tongue compression, displacement distance of the hyoid bone and cricoid cartilage plate, inter-common carotid artery distance, tracheal inner diameter change, and the area of the mask body at the upper edge, lower edge, and middle of the cricoid cartilage plate (via CT imaging)
Post-extubation complications | 24 hours after laryngeal mask extubation
  Evaluation of mucosal injury (visible bleeding during mask removal), hoarseness (patient-reported), sore throat (VAS 0-10, 0 = no pain, 10 = severe pain), and regurgitation (presence of gastric fluid in the oropharynx) at 24 hours post-extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Jiangling Wang, Dr, Principal Investigator — Zhejiang Cancer Hospital
Locations (2):
- China (2):
  - Ethics Committee of Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Jiangling Wang, Hangzhou, Zhejiang